CLINICAL TRIAL: NCT00627640
Title: A Phase III, Double-blind, Placebo-controlled, Randomised Trial to Determine the Efficacy and Safety of a Dose Range of 50 to 100 mg/Day of Safinamide, as add-on Therapy, in Subjects With Idiopathic Parkinson's Disease With Motor Fluctuations, Treated With a Stable Dose of Levodopa and Who May be Receiving Concomitant Treatment With Stable Doses of a Dopamine Agonist, an Anticholinergic and/or Amantadine
Brief Title: Safinamide in Idiopathic Parkinson's Disease (IPD) With Motor Fluctuations, as add-on to Levodopa
Acronym: SETTLE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Newron Pharmaceuticals SPA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27919; IND: 63,901; EudraCT Number: 2007-002964-90
Record Dates: First submitted 2008-02-13; First posted 2008-03-03 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2012-06

CONDITIONS: Idiopathic Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): 1 active (50 - 100 mg/day)
  Interventions: Drug: Safinimide 50-100 mg/day
- 2 (Placebo Comparator)
  Interventions: Drug: Matching Placebo

INTERVENTIONS:
Drug: Safinimide 50-100 mg/day — Safinamide, (S)-(+)-2-[4-(3-fluorobenzyloxy) benzylamino] propanamide methanesulfonate, is an a-aminoamide derivative
  Arms: 1
Drug: Matching Placebo — Matching Placebo
  Arms: 2

SUMMARY:
Parkinson's Disease is a major neurodegenerative disorder in which there is a progressive loss of dopamine-containing neurons. The understanding that PD is a syndrome of dopamine (DA) deficiency led to the introduction in the clinical practice of L-dopa, a precursor of DA that crosses the blood brain barrier, and also to the use of selective inhibitors of MAO-B, the major DA metabolising enzyme in man.

Safinamide is an inhibitor of MAO-B. This is a phase III trial to evaluate the efficacy and safety of safinamide (50 and 100 mg p.o. q.a.m.) compared to placebo as add-on therapy to a stable dose to levodopa in subjects with advance idiopathic Parkinson's Disease.

The principal efficacy measure is the increase in mean daily "on" time during the 18-hr diary recording period.

ELIGIBILITY:
Inclusion Criteria:

Male and female between the ages of 30 to 80 years with diagnosis of idiopathic Parkinson's Disease of more than 5 years duration, with a Hoehn and Yahr stage of I-IV during an "off" phase.

Be levodopa-responsive and have been receiving treatment with a stable dose of levodopa for at least 4 weeks.

Have motor fluctuations, with >1.5 hours "off" time during the day. Be able to maintain an accurate and complete diary (18-hour)

Exclusion Criteria:

Patients with medical conditions and/or taking concomitant medications that would have put them at risk, interfered with the study evaluations, or made them unable to complete the requirements of the study;.

Be in a late stage of Parkinson's Disease, and experiencing severe, disabling peak-dose or biphasic dyskinesia and/or unpredictable or widely swinging fluctuations in their symptoms.

Current diagnosis of substance abuse or history of alcohol or drug abuse in the past 3 months.

Have received treatment with safinamide previously. History of, or current depression psychosis (e.g. schizophrenia or psychotic depression) Evidence of dementia or cognitive dysfunction. History of allergic response to anticonvulsants, levodopa, or other anti-Parkinsonian agents.

Hypersensitivity or contraindications to MAO-B inhibitors. Ophthalmologic history including any of the following conditions: albino subjects, family history of hereditary retinal disease, progressive and/or severe diminution of visual acuity (i.e., 20/70), retinitis pigmentosa, retinal pigmentation due to any cause, any active retinopathy or ocular inflammation (uveitis), or diabetic retinopathy.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 549 (Actual)
Dates: Start 2009-02; Primary Completion 2012-01 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the change from baseline to W24 in daily "on" time ("on" time without dyskinesia plus "on" time with minor dyskinesia) | 24 weeks

SECONDARY OUTCOMES:
Evaluate the changes from baseline to W24 in Activities of Daily Living, cognition, dyskinesias, change in global clinical status, motor symptoms, motor fluctuations, change in levopoda dose and Health Related Quality of life | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Algirdas Kakarieka, MD, Study Director — Merck Serono S.A., Geneva
Locations (121):
- United States (28):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Barrow Neurological Institute, Phoenix, Arizona
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - San Francisco Clinical Research Center, San Francisco, California
  - Parkinson's Institute, Sunnyvale, California
  - Institute for Neurodegenerative Disorders, New Haven, Connecticut
  - Parkinson's Disease and Movement Disorder Center, Boca Raton, Florida
  - Neurologic Consultants P.A., Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - Parkinson's Disease Treatment Center of SW Florida, Port Charlotte, Florida
  - Neurology Clinical Research Inc., Sunrise, Florida
  - University Of South Florida Medical Center, Tampa, Florida
  - Wesley Woods Geriatric Center, Atlanta, Georgia
  - Columbus Research Institute, Columbus, Georgia
  - Northwestern University PD and Movement Disorders Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - Quest Research Institute, Bingham Farms, Michigan
  - Parkinson's Disease and Movement Disorder Center, Albany, New York
  - North Shore Medical Center, Manhasset, New York
  - Neurological Institute of New York, New York, New York
  - The Neurological Institute, Charlotte, North Carolina
  - Duke Movement Disorders Clinic, Durham, North Carolina
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor College of Medicine, Houston, Texas
- Australia (2):
  - Concord Repatriation General Hospital, Concord
  - Central Coast Neuroscience Research, East Gosford
- Austria (2):
  - Univ.Klinik Graz, Graz
  - Univ.Klinik Innsbruck, Innsbruck
- Belgium (6):
  - Cliniques Universitaires Saint-Luc, Brussels
  - U.Z Antwerpen, Edegem
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - ZNA Hoge Beuken, Hoboken
  - Heilig Hart Roeselare - Campus westlaan, Roeselare
  - AZ Sint-Augustinus, Wilrijk
- Canada (6):
  - Research Site, Halifax, Nova Scotia
  - Parkinson's and Neurodegenerative Disorders Clinic, Ottawa, Ontario
  - University Health Network -Toronto Western Hosp., Toronto, Ontario
  - Dynamic Clinical Research Group, Pointe-Claire, Quebec
  - King David, Halifax
  - Kingston General Hospital, Kingston
- Tartu University Hospital, Tartu, Estonia
- France (5):
  - CHU Hopital Gabriel Montpied, Clermont-Ferrand
  - CHU La Miletrie, Miletrie Poitiers
  - CHU Nantes Hôpital Laennec - CIC Neurologie, Nantes
  - CHU de Nimes, Hopital Caremeau, Nîmes
  - CIC-Hospital Purpan, Pavillon Riser Toulouse
- Germany (12):
  - Kliniken Beelitz GmbH, Beelitz-Heilstätten
  - Charité Campus Virchow Universitaetsmedizin Berlin, Berlin
  - Ehret Reinhard, Berlin
  - St. Joseph-Krankenhaus Berlin-Weißensee, Berlin
  - Universitaetsklinikum Goettingen, Göttingen
  - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Philipps-Universitaet Marburg, Marburg
  - Praxis Dipl med Bodenschatz, Mittweida
  - Neurologisches Krankenhaus Muenchen, München
  - Eberhard-Karls-Universität, Tübingen
  - Universitätsklinikum, Ulm
  - Deutsche Klinik fuer Diagnostik, Wiesbaden
- Hungary (12):
  - Clinexpert Kereskedelmi es Szolgaltato Kft., Budapest
  - Fov.Onk.Peterfy S.Utcai Korh.-Rend.Int es Baleseti Kozp., Budapest
  - Fővárosi Önkormányzat Nyírő Gyula Kórhaz Neurologiai Osztály, Budapest
  - Nyiro Gyula Korhaz, Budapest
  - Semmelweis Egyetem, Budapest
  - SOTE Neurlogia, Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum, Debrecen
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyetemi Oktato Korhaz, Miskolc
  - DE OEC Neurologiai Klinika, Móricz
  - Peterfy S. Utcai Korhaz, Peterfy Sandor
  - Sopron Medical Egeszsegugyi Szolgaltato Kft., Sopron
  - BAZ Country Hospital and Outpatient Clinic Dept. of Neurology Toxicology and Stroke, Szentpetri
- India (8):
  - Nizam's Institute of Medical Sciences, Hyderabad, Andh Prad
  - King George Hospital, Visakhapatnam, Andh Prad
  - M. S. Ramaiah Medical College and Hospital, Bangalore, Karna
  - All India Institute of Medical Sciences (AIIMS), New Delhi, National Capital Territory of Delhi
  - Mallikatta Neuro and Research Centre, Mangalore
  - BYL Nair Hospital ¬ TN Medical College, Mumbai Mahara
  - Brain & Mind Institute, Nagpur
  - Christian Medical College Hospital, Vellore
- Israel (6):
  - Barzilai Medical Center, Ashkelon
  - Rambam Health Care Campus, Haifa
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sieff Government Hospital, Safed
  - Sourasky Medical Center, Tel Aviv
- Malaysia (2):
  - Hospital Pulau Pinang, George Town
  - University of Malaya Medical Center, Kuala Lumpur
- Jeroen Bosch Ziekenhuis, 's-Hertogenbosch, Netherlands
- New Zealand (3):
  - Auckland City Hospital, Aucklan
  - Van der Veer Institute for Parkinson's & Brain Research, Christchurch
  - Waikato Hospital, Hamilton
- Slovakia (5):
  - MU Dr.Beata Dupejová neurologicka ambulancia s.r.o, Banská Bystrica
  - Poliklinika Tehelna, Bratislava
  - Vseobecna nemocnica s poliklinikou Levoca, Levoča
  - Fakultna nemocnica Trnava Interna klinika, Slovak Republic
  - Nestatne zdravotnicke zariadenie Neurologicka ambulancia, Slovak Republic
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University College of Medicine, Seoul
- Spain (4):
  - Policlinica Guipuzcoa, Donostia / San Sebastian
  - Fundacion Hospital de Alcorcon, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - HU Carlos Haya, Málaga
- Switzerland (2):
  - Inselspital Bern, Bern
  - Hopitaux Universitaires de Geneve - Hug, Geneva
- Taiwan (3):
  - Chang-Hua Christian Hospital, Chang-hua
  - Kaohsiung Veterans General Hospital, Kaohsiung City
  - Shin Kong Wu Ho-Su Memorial Hospital, Taipei
- Thailand (5):
  - King Chulalongkorn Memorial Hospital, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Rajavithi Hospital, Bangkok
  - Lampang Hospital, Lampang
  - Sappasithiprasong Hospital, Ubonratchathani
- United Kingdom (5):
  - Fylde Coast Hospital, Blackpool
  - Addenbrookes NHS Trust, Cambridge
  - Southern General Hospital, Glasgow
  - Royal Free Hospital, London
  - Clinical Ageing Research Unit, Newcastle upon Tyne

REFERENCES:
- [Derived] Cattaneo C, Kulisevsky J. The Effects of Safinamide in Chinese and Non-Chinese Patients with Parkinson's Disease. Adv Ther. 2024 Feb;41(2):638-648. doi: 10.1007/s12325-023-02736-2. Epub 2023 Dec 9. PMID 38070039
- [Derived] Schapira AH, Fox SH, Hauser RA, Jankovic J, Jost WH, Kenney C, Kulisevsky J, Pahwa R, Poewe W, Anand R. Assessment of Safety and Efficacy of Safinamide as a Levodopa Adjunct in Patients With Parkinson Disease and Motor Fluctuations: A Randomized Clinical Trial. JAMA Neurol. 2017 Feb 1;74(2):216-224. doi: 10.1001/jamaneurol.2016.4467. PMID 27942720